CLINICAL TRIAL: NCT07003139
Title: A Phase I/II Study to Evaluate Safety and Efficacy of the Boron Neutron Capture Therapy (BNCT) Using B10 L-BPA as Boron Carrier in Malignant Brain Tumors.
Brief Title: A Study of the Boron Neutron Capture Therapy (BNCT) Using B10 L-BPA in Malignant Brain Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Heron Neutron Medical Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH114-REC1-016
Record Dates: First submitted 2025-05-05; First posted 2025-06-04 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Malignant Brain Tumors
Keywords: L-4-(10B)Boronophenylalanine; (10B)-4-Borono-L-phenylalanine; BNCT; Malignant Brain Tumors; Boron Neutron Capture Therapy; Borofalan (10B)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Boron Neutron Capture Therapy (Experimental): Single arm treated by BNCT only
  Interventions: Drug: B10 L-BPA Injection

INTERVENTIONS:
Drug: B10 L-BPA Injection — The investigational product is B10 L-BPA Injection, is a boron-containing compound in which 10B replaces a position on L-phenylalanine at the para position with dihydroxyboron.

SUMMARY:
This Phase I/II study, titled 'A Phase I/II Study to Evaluate Safety and Efficacy of the Boron Neutron Capture Therapy (BNCT) using B10 L-BPA as Boron Carrier in Malignant Brain Tumors.', aims to assess the efficacy of B10 L-BPA with BNCT in patients with malignant brain tumors. The primary objective is to evaluate the safety and efficacy of BNCT with B10 L-BPA for malignant brain tumors treatment, using the Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) as the standard for assessment.

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years and older.
2. Patients with malignant brain tumors confirmed by histological and/or medical imaging, classified as WHO Grade 3 or 4 according to the World Health Organization of tumors of the central nervous system (CNS) classification, excluding those with histologically confirmed Grade 3 intracranial ependymoma, medulloblastoma, and primary CNS lymphoma.
3. There must be a time interval ≥ 3 months between prior radiation therapy and the scheduled BNCT.
4. There must be a time interval ≥ 1 month between receipt of antitumor drugs and the scheduled BNCT.
5. Within 4 weeks prior to the screening visit, measurable disease by magnetic resonance imaging (MRI) and/or computed tomography (CT) scan showing a volume ≦ 250 cm^3, longest dimension < 7 cm.
6. At least one measurable lesion that can be assessed by RECIST v1.1.
7. Eastern Cooperative Oncology Group (ECOG) Performance Score ≤ 2.
8. Life expectancy ≥ 3 months in the opinion of the investigator.
9. Adequate organ functions as defined below:

   * Hemoglobin ≥ 8.0 g/dL.
   * White blood cell (WBC) count ≥ 2.5 x 10^3/μL.
   * Neutrophil count ≥ 1.5 × 10^3/μL.
   * Platelet count ≥ 80 × 10^3/μL.
   * Aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN).
   * Alanine aminotransferase (ALT) ≤ 2.5 × ULN.
   * Serum creatinine ≤ 1.5 × ULN
   * Estimated glomerular filtration rate(eGFR) ≥ 15 mL / min / 1.73m^2
10. Female subjects with reproductive potential must have a negative result of serum pregnancy test at the screening visit and urine pregnancy test before the B10 L-BPA administration. However, if the subject has been menopausal for at least 2 years (more than 24 months since the last menstrual period) or uses surgical birth control, testing is not required.
11. Female subject with childbearing potential as well as male subject with reproductive potential must agree to refrain from unprotected sex and use 2 methods of highly effective contraception with their partner (e.g. barrier contraceptives [male condom, female condom, or diaphragm plus spermicide], intrauterine device, hormonal methods [hormone shot or injection, implants, combination oral contraceptives, or patches]) for ≥ 6 months after the BNCT until the end of this study.
12. Physically and mentally capable of participating in the study and willing to adhere to study procedures.
13. Provision of signed informed consent.

Exclusion Criteria:

1. Patients with malignant brain tumors complicated by any of the following conditions:

   * Extracranial metastases.
   * Multiple intracranial lesions on both sides.
2. The investigator assesses that the subject has concurrent infections or other malignant tumors and is not suitable to participate in the trial.
3. Patients with malignant brain tumors are considered eligible for standard surgical treatment that is effective against the tumor.
4. A time interval less than 3 months from previous radiation therapy for intracranial region.
5. A time interval less than 3 months from last brain surgery (excluding drainage procedures and biopsy) and less than 1 month from previous chemotherapy.
6. The adverse event of previous anti-tumor therapy were NCI-CTCAE V5.0 grade evaluation ≧ Class 3 (excluding alopecia and peripheral neuropathy).
7. Received or expect to receive any investigational drug, biologic or device within 1 month prior to the scheduled BNCT.
8. Patients receiving or expected to receive vascular endothelial growth factor inhibitors (except bevacizumab) or live attenuated vaccines within 1 month prior to the scheduled BNCT.
9. Patients received major surgery within 1 month prior to the scheduled BNCT or are still recovering from a previous surgery. The investigator will evaluate the subject's condition when the subject receives major surgery. Major surgery is defined as procedure that requires general anaesthesia and/or anticipated hospitalization longer than 24 hours, with significant risk of blood loss or complications. Examples include heart surgery, organ transplants, and prolonged operations such as certain back surgeries. Procedures such as stent implantation, biopsy, endoscopy, and day surgery are excluded.
10. Patients who had radiation myelitits or radiation necrosis of the brain/brain stem.
11. Patient who is prone to vascular rupture during the trial as assessed by the investigator. The Patient will be eligible for the study if they have undergone stent implantation and obtained consent from the investigator.
12. Patients with severe congestive heart failure or renal failure, as well as myocardial infarction, unstable angina, or poorly controlled arrhythmia within 6 months prior to the scheduled BNCT.
13. Severe comorbidities, including but not limited to poorly controlled epilepsy, poorly controlled diabetes mellitus, poorly controlled hypertension; chronic lung diseases (e.g., obstructive pneumonia, interstitial pneumonia, pulmonary fibrosis, and severe emphysema); kidney diseases (e.g., chronic renal failure, acute renal failure and nephrotic syndrome); cardiac diseases (e.g., New York Heart Association [NYHA] Functional Classification Class III or IV); phenylketonuria; and/or other severe conditions in the opinion of the investigator.
14. Suspected or known hypersensitivity (including allergy) to boron or any component of the study drug or contrast media.
15. Subject with hereditary fructose intolerance.
16. With a cardiac pacemaker or will interfere with MRI-based or CT-based dose-planning or tumor response evaluation.
17. Restless subjects who are unable to lie or sit in a cast for more than 30 minutes.
18. Any medical or psychiatric conditions that, in the opinion of the investigator, may interfere with optimal participation in the study or place the subject at increased risk of adverse events (AEs).
19. Female subject who is planning to be pregnant or lactating during the study period.
20. Subject who is considered unfit to participate in the clinical study as assessed by the investigator.
21. Subject who has received prior BNCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety of BNCT using B10 L-BPA in treating malignant brain tumors | 6 months
  Safety will be assessed by monitoring the occurrence, severity, and relationship of treatment-emergent adverse events (TEAEs), including serious adverse events and events leading to permanent discontinuation of therapy, according to protocol definitions and CTCAE v5.0.
Efficacy of BNCT using B10 L-BPA in treating malignant brain tumors | 6 months
  Efficacy of BNCT with B10 L-BPA for treating malignant brain tumors will be assessed by the percentage of subjects achieving complete response (CR) and partial response (PR). Tumor response will be evaluated using RECIST v1.1 criteria via high-resolution CT or MRI.

SECONDARY OUTCOMES:
Progression-free survival | 6 months
  PFS is defined as the time from receiving the B10 L-BPA-based BNCT until progressive disease (PD) or death from any cause, whenever comes the first. PFS is evaluated by imaging according to the RECIST v1.1 criteria.
Change in Quality of Life as Measured by the EORTC QLQ-C30 Questionnaire | 6 months
  The EORTC QLQ-C30 is a validated questionnaire that evaluates cancer patients' quality of life through functional, symptom, and global health scales. It primarily using a 4-point scale (1='Not at All' to 4='Very Much'), and a 7-point scale for two items, where higher scores indicate more symptoms.
Change in Quality of Life as Measured by the EORTC QLQ-BN20 Questionnaire | 6 months
  The EORTC QLQ-BN20 is a validated module for brain tumor patients that assesses disease- and treatment-specific symptoms such as motor dysfunction, communication issues, and visual or cognitive changes. It uses a 4-point scale (1 = "Not at All" to 4 = "Very Much"), where higher scores indicate more severe symptoms.

OTHER OUTCOMES:
The population of circulating immune cells | 6 months
  Blood samples will be collected to assess MDSCs, T cells and IL-1β at multiple time points: before and after BNCT. This approach aims to clarify whether the levels of circulating immune cells could serve as prognostic indicators for BNCT treatment outcomes.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - China Medical University Hsinchu Hospital, Hsinchu
  - China Medical University Hospital, Taichung